CLINICAL TRIAL: NCT02999971
Title: Effects of an Aquatic Circuit Class Therapy Program Versus a Land Circuit Class Therapy Program in Patients Who Suffered a Stroke
Brief Title: Effects of an Aquatic Therapy Program Versus a Land Program in Patients Who Suffered a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, IRENE PEGITO PEREZ, Physiotherapy degree, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCoruna
Record Dates: First submitted 2016-12-18; First posted 2016-12-21 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Hydrotherapy
Keywords: circuit class therapy; ICF model; aquatic therapy; neuro-rehabilitation
MeSH Terms: conditions — Stroke | interventions — Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- circuit class therapy in water (Experimental): CCT on water. The intervention developed in this study will be through the realization of an exercise program in circuit (CCT). One of the groups will receive treatment in the water (intervention group), and the other on land (control group). In both groups, the intervention will be a 7-week class therapy, 3-times weekly, giving a total of 20 sessions.
  Interventions: Other: circuit class therapy in water
- circuit class therapy on land (Experimental): CCT on land. The intervention developed in this study will be through the realization of an exercise program in circuit (CCT). One of the groups will receive treatment in the water (intervention group), and the other on land (control group). In both groups, the intervention will be a 7-week class therapy, 3-times weekly, giving a total of 20 sessions.
  Interventions: Other: circuit class therapy on land

INTERVENTIONS:
Other: circuit class therapy in water — The circuit, the main part of the session, include a series of 10 different workstations, arranged to progress in complexity, in order to work several segments of the body, oriented towards a functional recovery objective. These stations will be made up of task-specific activities for gait, balance and dexterity. Time in each workstation will be 5 minutes divided as follows: 4 minutes work period and 1 minute rest period, of these, last 30 seconds will be change period for crossing from one workstation to the next. After 50 minutes, each patient will have covered the 10 workstations, thus working in all of the objectives pursued in the realization on this CCT: gait, balance and dexterity.
  Arms: circuit class therapy in water
Other: circuit class therapy on land — The circuit, the main part of the session, include a series of 10 different workstations, arranged to progress in complexity, in order to work several segments of the body, oriented towards a functional recovery objective. These stations will be made up of task-specific activities for gait, balance and dexterity. Time in each workstation will be 5 minutes divided as follows: 4 minutes work period and 1 minute rest period, of these, last 30 seconds will be change period for crossing from one workstation to the next. After 50 minutes, each patient will have covered the 10 workstations, thus working in all of the objectives pursued in the realization on this CCT: gait, balance and dexterity.
  Arms: circuit class therapy on land

SUMMARY:
The objective of this study is to investigate the relative effectiveness of CCT on water versus on land in stroke patients. Additionally, the study will to determine if there are differences in the results obtained, between two CCT programs in the following parameters: gait, balance and dexterity

DETAILED DESCRIPTION:
This study is a randomized controlled trial of the effectiveness of a structured CCT program in water versus a structured CCT program on land in the rehabilitation of stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of stroke (ischemic or hemorrhagic) onset ≤ 3 years; with hemiparesis secondary;
* age ≥18 to ≤ 90;
* provide a written informed consent;
* able to walk for at least 10 m without assistance

Exclusion Criteria:

* patients with uncontrolled or risky conditions (acute myocardial infarction, arrhythmia, heart failure, uncontrolled hypertension or unstable cardiovascular state);
* with infectious diseases, ulcers or urinary and / or faecal incontinence;
* additional neurological and / or orthopedic deficits that alter ambulation;
* unable to follow treatment (cognitive, visual ...).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
10 meters walk test | 60 seconds

SECONDARY OUTCOMES:
Test Up & Go | 5 minutes
Berg Balance Scale (BBS) | 20 minutes
Romberg Test | 1 minute
Fugl-Meyer Assessment | 15 minutes
Functional Reach Test (FRT) | 10 minutes
Box and block test | 5 minutes
Self-efficacy Scale | 5 minutes
Activities-Specific Balance Confidence Scale (ABC) | 10 minutes

IPD SHARING:
Plan to Share IPD: No